CLINICAL TRIAL: NCT00569972
Title: PD 0200390 Dose Ranging Trial: A Randomized, Double Blind, Parallel Group, Placebo Controlled, Multicenter Outpatient Trial Of PD 0200390 In Adults With Primary Insomnia
Brief Title: A Randomized, Double Blind, Parallel Group, Placebo Controlled, Multicenter Outpatient Trial Of PD 0200390 In Adults With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4251037
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — (1-aminomethyl-3,4-dimethylcyclopentyl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 15 mg PD 0200390 (Experimental)
  Interventions: Drug: PD 0200390
- 30 mg PD 0200390 (Experimental)
  Interventions: Drug: PD 0200390
- 45 mg PD 0200390 (Experimental)
  Interventions: Drug: PD 0200390
- 60 mg PD 0200390 (Experimental)
  Interventions: Drug: PD 0200390
- Placebo PD 0200390 (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PD 0200390 — Capsules, 15 mg, 3 capsules each night before bedtime, Duration - Visit 3-7 for 28 days
  Arms: 15 mg PD 0200390
Drug: PD 0200390 — Capsules, 30 mg, 3 capsules each night before bedtime; Duration - Visit 3-7 for 28 days
  Arms: 30 mg PD 0200390
Drug: PD 0200390 — Capsules, 45 mg, 3 capsules each night before bedtime, Duration- Visit 3-7 for 28 days
  Arms: 45 mg PD 0200390
Drug: PD 0200390 — Capsules, 60 mg, 3 capsules each night before bedtime, Duration - Visit 3-7 for 28 days
  Arms: 60 mg PD 0200390
Drug: Placebo — Matched oral placebo for weeks 2-7.
  Arms: Placebo PD 0200390

SUMMARY:
To demonstrate efficacy and characterize the dose response relationship of PD 0200390 on subjective wake after sleep onset in subjects with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* 3 month history of primary insomnia;
* 18 to 64 years
* For the last 3 months-regularly awake unrefreshed and unrestored
* Difficulty initiating and maintaining sleep for at least 3 nights/week for the past month (difficulty falling asleep, difficulty staying asleep, early awakening)

Exclusion Criteria:

* Any history of an Axis 1 psychiatric diagnosis;
* History or presence of any breathing related sleep disorder;
* History or presence of any medical or neurological condition that could interfere with sleep
* Use of alcohol as a sleep aid or more than 2 standard drinks consumed per day or more than 14 consumed per week

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 682 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate efficacy and characterize the dose response relationship of PD 0200390 on subjective wake after sleep onset in subjects with primary insomnia. | Weekly

SECONDARY OUTCOMES:
To characterize the dose response relationship of PD 0200390 on functional outcome measures in subjects with primary insomnia. | Weekly
To characterize the exposure response relationship of safety & efficacy parameters following administration of PD 0200390 in subjects with primary insomnia. | Weekly
To investigate the potential for rebound insomnia and withdrawal effects after discontinuation of PD 0200390 in subjects with primary insomnia. | Weekly
To characterize the dose response relationship of PD 0200390 on subjective assessments of latency to sleep onset (LSO), number of awakenings after sleep onset (sNAASO) and total sleep time (sTST) in subjects with primary insomnia. | Weekly
To investigate the safety and tolerability of PD 0200390 administered once daily before bedtime in subjects with primary insomnia. | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (70):
- United States (60):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Sherman Oaks, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Spring Hill, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Gainsville, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Mount Sterlingg, Kentucky
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Saint Clair Shores, Michigan
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Canada (10):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Sydney, Nova Scotia
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Etobicoke, Ontario
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Parry Sound, Ontario
  - Pfizer Investigational Site, Toronto, Ontario